CLINICAL TRIAL: NCT02262130
Title: Phase 2 Multicentric Study Evaluating the Efficacy of Omalizumab in Idiopathic Severe and Refractory Solar Urticaria
Brief Title: Omalizumab in Severe and Refractory Solar Urticaria
Acronym: XOLUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2013/209
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Solar Urticaria
Keywords: Omalizumab; Efficacy; Safety
MeSH Terms: conditions — Urticaria, Solar | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omalizumab (Experimental): Omalizumab 300 mg W0, W4 and W8
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
Solar urticaria is a rare disease, with a usual favourable outcome with photoprotection and with anti H1 histamines. Nevertheless, some cases can be severe and refractory to this usual treatment, leading to a large impact on quality of life. New treatment options are warranted. The investigators aim to test the efficacy and the safety of omalizumab, an anti-IgE antibody recently approved in chronic spontaneous urticaria, in this setting.

DETAILED DESCRIPTION:
This is an open-labelled multicentric phase II study testing the efficacy and the safety of omalizumab 300 mg (W0, W4 and W8) in patients affected with severe and refractory solar urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years,
* Appearance of wheals within 15 min after sun exposure and lasting < 2 hr in the shade,
* Wheals reproducible with phototesting: appearance after exposure to UVB, UVA or visible light less than 30 min after exposure and lasting < 2 hr,
* Severity criteria:

  * Very large effect on quality of life, with Dermatology Life Quality Index (DLQI) > 10, and
  * At least 1 of the following: involvement of the face, per annual eruption, extension of wheals on the non-photoexposed skin, SU triggered by artificial light, SU flares accompanied by bronchospasm or syncope.
* Refractory criteria:

  * Resistance to photoprotection with sunscreen with sun protection factor ≥ 50, and
  * Resistance to administration of an association of 2 different antihistamines during 3 months or to photodesensitization.

Exclusion Criteria:

* Contra indication to omalizumab
* Previous treatment with omalizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuelle Viguier, MD, PhD, Principal Investigator — Assistance Publique-Hôpitaux de Paris, Université Paris 7; François AUBIN, Prof., Principal Investigator — Centre hospitalier régional universitaire de Besançon
Locations (13):
- France (13):
  - CHU de Angers, Angers
  - Dermatology department, Centre Hospitalier Régional Universitaire, Besançon
  - CHU de Caen, Caen
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - Dermatology department, Hôpital Saint-Louis, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: Omalizumab 300 mg W0, W4 and W8
  Omalizumab
Period: Overall Study
Arm/Group | Omalizumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omalizumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Remission of Solar Urticaria Under Experimental Conditions (Phototesting)
Description: Proportion of patients with minimal urticarial dose (MUD) increased compared to baseline, under experimental conditions (assessed by phototesting).
  A small area of skin is exposed to increasing UVA doses with a solar simulator until an allergic reaction appears. The lower UVA dose triggering the urticaria is the MUD.
Time Frame: 4 weeks after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab
Number analyzed (Participants) | 10
Participants | 2

2. Secondary Outcome: Proportion of Patients for Whom the Treatment Allowed Achieving Dermatology Life Quality Index< 6
Description: Proportion of patients for whom the treatment with omalizumab allowed achieving DLQI < 6.
  The index extends from 0 to 30: 0 - 1 = no effect at all on patient's life / 2 - 5 = small effect on patient's life / 6 - 10 = moderate effect on patient's life / 11 - 20 = very large effect on patient's life / 21 - 30 = extremely large effect on patient's life
Time Frame: 4 and 12 weeks after the end of treatment
Population: 1 patient withdrawn between week 12 and week 20 (discontinuation)
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab
Number analyzed (Participants) | 10
Participants
  4 weeks after the end of treatment | 4
  12 weeks after the end of treatment: number analyzed (Participants) | 9
  12 weeks after the end of treatment | 1

3. Secondary Outcome: Proportion of Patients With Solar Urticaria Remission Under Experimental Conditions (Phototesting)
Description: as for outcome 1
Time Frame: 12 weeks after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Proportion of Patients Achieving 50% Improvement in Solar Urticaria Intensity
Description: Proportion of patients achieving 50% improvement in solar urticaria intensity, compared to baseline, assessed by Visual Analogic Scale (scale extending from 0 to 10)
Time Frame: 4 and 12 weeks after the end of treatment
Population: 1 patient withdrawn between week 12 and week 20 (discontinuation)
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab
Number analyzed (Participants) | 10
Participants
  4 weeks after the end of treatment | 4
  12 weeks after the end of treatment: number analyzed (Participants) | 9
  12 weeks after the end of treatment | 0

5. Secondary Outcome: Proportion of Patients Achieving Clinical Remission of Solar Urticaria
Description: Proportion of patients showing no or less clinical signs or solar urticaria compared to baseline, under experimental conditions
Time Frame: 4 and 12 weeks after the end of treatment
Population: 1 patient withdrawn between week 12 and week 20 (discontinuation)
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab
Number analyzed (Participants) | 10
Participants
  4 weeks after the end of treatment | 3
  12 weeks after the end of treatment: number analyzed (Participants) | 9
  12 weeks after the end of treatment | 1

ADVERSE EVENTS:
Arm/Group | Omalizumab
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=10)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Patient treated from 12th November 2014 to 17th June 2015. A positive pregnancy test was performed in September 2015 with echographic confirmation.
Cholecystectomy (Hepatobiliary disorders) | 1 (1) — Gallbladder removal
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=10)
Headache (Nervous system disorders) | 6 (37)
Nausea (Gastrointestinal disorders) | 4 (21)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (16)
Asthenia (General disorders) | 3 (5)
Injection site reaction (General disorders) | 2 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Influenza (Infections and infestations) | 2 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Zona (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Faintness (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iron deficiency (Investigations) | 1 (1)
Solar urticaria relapse (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No